CLINICAL TRIAL: NCT02542098
Title: A Phase 2B, Open-label, Multicenter Study Evaluating the Safety, Pharmacokinetics, and Effectiveness of Hydrocodone Bitartrate Extended-Release Tablets (HYD) in Children, Aged 12 to 17 Years Inclusive, With Moderate to Severe Malignant and/or Nonmalignant Pain Requiring Around-the-Clock Opioid Analgesics
Brief Title: Safety, Pharmacokinetics (PK), and Effectiveness of Hydrocodone Bitartrate (HYD) Extended-Release Tablets in Children
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been updated with a new protocol number
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYD4002
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HYD 20 - 120 mg (Experimental): Hydrocodone bitartrate 20 mg to 120 mg extended-release tablets administered orally every 24 hours
  Interventions: Drug: HYD tablets

INTERVENTIONS:
Drug: HYD tablets — Hydrocodone bitartrate 20 mg to 120 mg extended-release tablets.
  Other Names: Hysingla® ER

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and effectiveness of Hydrocodone Bitartrate (HYD) tablets in children with moderate to severe pain requiring around-the-clock opioid analgesics.

ELIGIBILITY:
Inclusion Criteria include:

1. Males and females, aged 12 to 17 years, with pain severe enough to require daily, around-the-clock opioid treatment at a dose equivalent to at least 20 mg daily of hydrocodone for at least 2 weeks.
2. Patients must have stable vital signs and hemoglobin oxygen saturation, eg, measured by pulse oximetry (SpO2).
3. Patients must be willing and able to swallow medicinal tablets.
4. Female patients of childbearing potential must have a negative pregnancy test within 24 hours prior to the start of study drug treatment.
5. Female patients who are sexually active must be using (and continue using throughout the study) an acceptable method of birth control, per investigator's discretion.
6. Patients and patient's parent/caregiver must be compliant with the protocol, ie, must be able to perform study assessments and understand and complete the age-appropriate scale to rate pain intensity.
7. Patients must not have a cognitive developmental delay or any other condition that would preclude them from completing the age-appropriate pain scale.

Exclusion Criteria include:

1. Patients who require a starting total daily dose of HYD > 120 mg.
2. Patients who have had surgery within 72 hours prior to the start of study drug treatment.
3. Patients who have any planned surgery during the study will be excluded.
4. Female patients who are pregnant or lactating.
5. Patients who are allergic to hydrocodone or any other component of HYD or have a history of allergies to other opioids.
6. Patients who receive or are expected to receive an investigational drug/therapy during the study drug treatment or follow-up period.
7. Patients who are anticipated to receive any hydrocodone- or hydromorphone-containing products (other than study drug) during the study or 3 days prior to initiation of treatment with study drug.
8. Patients with a history of alcohol, medication, or illicit drug abuse or addiction and/or opioid abuse or addiction at any time.
9. Patients with contraindication to blood sampling.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
The number of participants with adverse events as a measure of safety | Up to 4 weeks (during the study) and 7-10 days poststudy (safety follow-up assessment).
Pharmacokinetic analysis to characterize the apparent volume of distribution (Vc/F) of hydrocodone following oral administration | Day 1, End of week 2, End of week 4
Pharmacokinetic analysis to characterize the apparent oral clearance (CL/F) of hydrocodone following oral administration | Day 1, End of week 2, End of week 4

SECONDARY OUTCOMES:
"Pain Right Now" Assessment by Patients using 100-mm visual analog scale (VAS) | Day 1 up to week 4
Parent/ Caregiver-Assessed Global Impression of Change (PGIC) | Week 4 / end of treatment